CLINICAL TRIAL: NCT06455306
Title: Erythritol Air Polishing in Mucositis Treatment: A Randomized Controlled Trial
Brief Title: Erythritol Air Polishing in Mucositis Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Orlando Martins, Visiting Assistant Professor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mucositis_Erythritol
Record Dates: First submitted 2024-05-18; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Peri-implant Mucositis
Keywords: peri-implant mucositis; erythritol powder air-polishing; non-surgical treatment
MeSH Terms: interventions — Erythritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group Erythritol Monthly Applications (Experimental): Patients will receive monthly applications (months 0, 1, and 2) of treatment with an air-polishing device with erythritol, along with oral hygiene instructions
  Interventions: Procedure: Air-polishing with erythritol at different time points
- Control group (No Intervention): Patients will receive only oral hygiene instructions
- Test Group Erythritol Single Application (Experimental): Patients will receive a single application of treatment with an air-polishing device with erythritol, in addition to oral hygiene instructions
  Interventions: Procedure: Single Air-polishing with erythritol

INTERVENTIONS:
Procedure: Air-polishing with erythritol at different time points — The air-polishing device will be inserted into each site of the peri-implant pocket at an angle ranging from 60 to 90 degrees, and each surface will be debrided for 5 seconds using erythritol powder (AIRFLOW Powder PERIO; EMS). In this group this procedure will be done ate baseline, 1 month and 2 months
  Arms: Test Group Erythritol Monthly Applications
Procedure: Single Air-polishing with erythritol — The air-polishing device will be inserted into each site of the peri-implant pocket at an angle ranging from 60 to 90 degrees, and each surface will be debrided for 5 seconds using erythritol powder (AIRFLOW Powder PERIO; EMS). In this group this procedure will be done ate baseline only.
  Arms: Test Group Erythritol Single Application

SUMMARY:
This study aimed to evaluate the effectiveness of air polishing systems compared to the exclusive use of oral hygiene instruction in the treatment of peri-implant mucositis

DETAILED DESCRIPTION:
The study will include individuals aged 18 to 80 who have at least one implant and exhibit peri-implant mucositis, as defined by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions.

Participants will be selected from those attending Periodontology, Oral Surgery, and Oral Medicine consultations at the dental medicine clinic of the University Hospital Center of the University of Coimbra (CHUC). After confirming the inclusion and exclusion criteria, patients will be invited to participate in the study, and if they agree to participate, they will sign an Informed Consent Form.

The study is conducted as a parallel-design clinical trial, and each participant will be randomly allocated to one of three groups: Test 1 (T1), Test 2 (T2), or Control (C).

Group T1 will consist of patients receiving a single application of treatment with an air-polishing device with erythritol, in addition to oral hygiene instructions (OHI). Group T2 will consist of patients receiving monthly applications (months 0, 1, and 2) of treatment with an air-polishing device with erythritol, along with OHI. Group C will consist of patients receiving only OHI. The treatments and OHI will be performed by an experienced periodontist who is different from the one collecting clinical, radiographic, and PICF data.

The clinical examination that will be performed at baseline, 3 and 6 months after baseline includes a periodontal chart at six sites per each tooth and/or included implant.

In addition, collection of peri-implant crevicular fluid (PICF) will be done to evaluate a panel of biomarkers. Samples will be collected from two locations around each implant, isolated with cotton rolls and dried. Using the filter paper technique, a strip of standard length and height filter paper (Periopaper, Pro Flow, New York, USA) will be inserted into the peri-implant sulcus and left in place for 30 seconds. Samples will be placed in plastic centrifuge tubes and kept on ice until they are frozen (-80°C) in the laboratory of the Clinical Pathology Service at CHUC. Sampling should be performed prior to peri-implant clinical examination and after gentle removal of supra-gingival plaque. Biochemical analysis will be conducted using Luminex to evaluate the inflammatory pattern through the use of a panel of biomarkers.

Schedule of appointments by Group:

* Group T1: Month 0 appointment (collection of clinical data, X-rays, and Peri-implant crevicular fluid (PICF); OHI + treatment); Month 3 appointment (collection of clinical data and PICF); Month 6 appointment (collection of clinical data, X-rays, and PICF).
* Group T2: Month 0 appointment (collection of clinical data, X-rays, and PICF; OHI + treatment); Month 1 appointment (OHI + treatment); Month 2 appointment (OHI + treatment); Month 3 appointment (collection of clinical data and PICF); Month 6 appointment (collection of clinical data, X-rays, and PICF).
* Group C: Month 0 appointment (collection of clinical data, X-rays, and PICF; OHI); Month 3 appointment (collection of clinical data and PICF); Month 6 appointment (collection of clinical data, X-rays, and PICF).

ELIGIBILITY:
Inclusion Criteria:

* Adults with at least one implant in function for a minimum of one year affected by peri-implant mucositis.

Exclusion Criteria:

1. Pregnant or lactating women
2. patients unable to understand the treatment protocol and sign informed consent and/or patients younger than 18 years old,
3. medical conditions that prevents an oral examination,
4. incapability to perform oral hygiene measures due to physical or mental disorders,
5. patients with uncontrolled systemic diseases or neoplasms, infection with HIV or hepatitis, cardiovascular disease, blood disorders (e.g. coagulation disorders) and severe osteoporosis,
6. patients who have received systemic antibiotics, corticosteroids, or immunosuppressive therapy within 3 months before periodontal evaluation (baseline), as well as those who chronically use nonsteroidal anti-inflammatory drugs, require antibiotic coverage for dental procedures, and those who are undergoing chronic treatment with medications known to affect periodontal health (such as phenytoin or cyclosporine),
7. alcohol or drug addiction
8. implants with mobility and/or occlusal overload.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Bleeding on Probing compared to baseline | Baseline, 3 months and 6 months
  Bleeding on Probing (BoP) will be evaluated according to the modified bleeding index (0-no BoP; 1- punctiform drop of bleed; 2- confluent red continuous line formed through the sulcus; 3-heavy/profuse), for each site

SECONDARY OUTCOMES:
Probing Pocket Depth | Baseline, 3 months and 6 months
  Measured in mm from the mucosal margin to most apical point of the pocket
Plaque index (PI) | Baseline, 3 months and 6 months
  assessed dichotomously as the presence or absence of plaque along the mucosal/gingival margin
Gingival Recession | Baseline, 3 months and 6 months
  Distance, measured in mm from the cementoenamel junction to the gingival margin
Radiographic bone level | Baseline, 3 months and 6 months
  calculated as the difference between the marginal bone levels assessed at follow-up visits and the ones assessed in the baseline
Biochemical outcomes | Baseline, 3 months and 6 months
  Peri-implant crevicular fluid (PICF) analysis: a collection of PICF samples will be done to evaluate a panel of biomarkers (IL-4, IL-6, IL-10, IL-1B)
Complete Disease Resolution | 3 months and 6 months
  Total Absence of bleeding on probing and deep probing pocket depths on the implant site
Keratinized Tissue | Baseline, 3 months and 6 months
  Measure in mm in the vestibular site
Prosthetic Margin Level | Baseline, 3 months and 6 months
  Level of the prosthetic implant connection regarding the gingival margin

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Martins, Study Director — Visiting Assistant Professor
Locations (1):
- University of Coimbra, Coimbra, Portugal

REFERENCES:
- [Background] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Background] Renvert S, Persson GR, Pirih FQ, Camargo PM. Peri-implant health, peri-implant mucositis, and peri-implantitis: Case definitions and diagnostic considerations. J Clin Periodontol. 2018 Jun;45 Suppl 20:S278-S285. doi: 10.1111/jcpe.12956. PMID 29926496
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Lee CT, Huang YW, Zhu L, Weltman R. Prevalences of peri-implantitis and peri-implant mucositis: systematic review and meta-analysis. J Dent. 2017 Jul;62:1-12. doi: 10.1016/j.jdent.2017.04.011. Epub 2017 May 3. PMID 28478213
- [Background] Herrera D, Berglundh T, Schwarz F, Chapple I, Jepsen S, Sculean A, Kebschull M, Papapanou PN, Tonetti MS, Sanz M; EFP workshop participants and methodological consultant. Prevention and treatment of peri-implant diseases-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2023 Jun;50 Suppl 26:4-76. doi: 10.1111/jcpe.13823. Epub 2023 Jun 4. PMID 37271498
- [Background] Romandini M, Lima C, Pedrinaci I, Araoz A, Soldini MC, Sanz M. Prevalence and risk/protective indicators of peri-implant diseases: A university-representative cross-sectional study. Clin Oral Implants Res. 2021 Jan;32(1):112-122. doi: 10.1111/clr.13684. Epub 2020 Dec 29. PMID 33210772
- [Background] Verket A, Koldsland OC, Bunaes D, Lie SA, Romandini M. Non-surgical therapy of peri-implant mucositis-Mechanical/physical approaches: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:135-145. doi: 10.1111/jcpe.13789. Epub 2023 Feb 28. PMID 36802083